CLINICAL TRIAL: NCT02970175
Title: Interest of in Situ Terlipressin Administration Before the Realisation of Bronchial Biopsy
Acronym: TERLAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014/0212/HP
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Bronchial Endoscopy
Keywords: Terlipressin
MeSH Terms: interventions — Chorionic Villi Sampling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchoscopy with terlipressin administration (Experimental): Patients undergoing a bronchoscopy under local anesthesia for biopsy sampling of endobronchial lesions. Bronchoscopy will be done with terlipressin administration
  Interventions: Drug: Terlipressin administration; Procedure: bronchoscopy under local anesthesia; Procedure: Biopsy sampling
- Bronchoscopy without terlipressin administration (Placebo Comparator): Patients undergoing a bronchoscopy under local anesthesia for biopsy sampling of endobronchial lesions. Bronchoscopy will be done without terlipressin administration
  Interventions: Procedure: bronchoscopy under local anesthesia; Procedure: Biopsy sampling

INTERVENTIONS:
Drug: Terlipressin administration — Patients undergoing a bronchoscopy under local anesthesia for biopsy sampling of endobronchial lesions. Bronchoscopy will be done with terlipressin administration
  Arms: Bronchoscopy with terlipressin administration
Procedure: bronchoscopy under local anesthesia — Patients undergoing a bronchoscopy under local anesthesia for biopsy sampling of endobronchial lesions. Bronchoscopy will be done with terlipressin administration
Procedure: Biopsy sampling — Patients undergoing a bronchoscopy under local anesthesia for biopsy sampling of endobronchial lesions. Bronchoscopy will be done with terlipressin administration

SUMMARY:
The diagnostic yield of flexible bronchoscopy for the diagnosis of lung cancer depends on the location and the histological type of the lesion, as well as on the number of biopsy samples performed. The increasing number of sampling is also important to provide material for molecular assessment of lung cancer. The French National Institute for Cancer recommends a number of 5 biopsies in order to reach a diagnostic yield of 88%. However, as increasing the number of bronchial biopsies comes with a higher risk of bleeding, the management of endobronchial bleeding may be determinant for the diagnostic yield.

The most recent recommendations of the British Thoracic Society for the management of bronchial bleeding, after bronchial or transbronchial biopsy, are to inject 5 to 10 mL of 1/10000 diluted adrenalin, or cold saline serum (04°C.). The French guidelines also include the use of endobronchial terlipressin, which has local vasoconstriction effect. After endobronchial administration of terlipressin, plasmatic concentrations are low, and are not clinically relevant.

The hypothesis of this clinical trial is that endobronchial instillation of terlipressin before sampling endobronchial tumor will limit the endobronchial bleeding and allow to increase the number of biopsies performed and, eventually, the diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Patients scheduled to undergo bronchoscopy, presenting a suspicious radiographic lesion and a lesion proximal tumor pace viewable in white light endoscopy and without pathologic diagnosis
* Patient having read and understood the information letter and signed the consent form
* Effective contraception in women of childbearing age

Exclusion Criteria:

* Patients with contraindication to the use of terlipressin:
* septic shock ,
* Hypersensitivity to terlipressin or the excipients or by whom use the product is not recommended:
* Recent history (<3 months) of acute coronary syndrome (including myocardial infarction) or unbalanced coronary insufficiency, or disorders of the ventricular heart rate.
* severe uncontrolled hypertension,
* cerebrovascular insufficiency and ischemic stroke of recent origin (<3 months).
* severe arterial occlusive lower extremities,
* severe chronic renal impairment (GFR <20 ml / min).
* Patients receiving uninterrupted antiplatelet therapy during 5 days before endoscopy (7 days for Clopidogrel Related), including low dose aspirin (≤ 75 mg / day).
* Patients receiving anticoagulant therapy:
* Unfractionated heparin within 12 hours before endoscopy.
* low molecular weight heparin within 24 hours before endoscopy.
* Patients with bleeding disorders defined by TP below 70% or TCA ratio patient / control greater than 1.3.
* Patients with thrombocytopenia less than 100 g / L.
* Subjects misunderstanding of spoken and written French
* Person under guardianship or deprived of liberty by judicial or administrative decision (under Article L1121-6 and L1121-8 of Public Health Code
* Pregnant or lactating women, premenopausal women without adequate contraception
* Patient participating in other drug testing or participating in another drug test in the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Number of biopsy realized during the endoscopy | Day 1
  The number of biopsy by endoscopy realized into each group will be calculated

SECONDARY OUTCOMES:
Number of biopsy allowing an histological diagnosis | Day 1
  The number of biopsy allowing an histological diagnosis into each group will be calculated
Number of adverse events due to terlipressin administration | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu SALAUN, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No